CLINICAL TRIAL: NCT01565499
Title: Phase II, Open-label, Non-randomized Study of Nab-paclitaxel for the Neoadjuvant Treatment of Patients With Stage II and III Luminal Breast Cancer
Brief Title: Neoadjuvant Treatment With Nab-paclitaxel for Patients With Stage II and III Luminal Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM/2011-02
Record Dates: First submitted 2012-03-22; First posted 2012-03-28 (Estimated); Results first posted 2020-11-18 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: Neoadjuvant nab-paclitaxel luminal breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nab-Paclitaxel (Experimental): The patients will be included to receive 3 weekly nab-paclitaxel doses of 150 mg/m2 with one week of rest for 4 cycles.
  Interventions: Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Nab-paclitaxel
  Other Names: Abraxane

SUMMARY:
Multicenter, open label, non-randomized phase 2 trial to evaluate the efficacy and safety of nab-paclitaxel in the neoadjuvant treatment of ER positive human epidermal growth factor receptor 2 (HER2) negative patients amenable to receive neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
The primary objective of the trial is to determine the percentage of patients with poor response [residual cancer burden III (RCB-III) rate] in contrast to good response [residual cancer burden 0/I RCB-0/1] measured by the Symmans criteria [20] at surgery, in patients with stage II-III luminal breast cancer treated with neoadjuvant nab-paclitaxel.

The primary endpoint of the study is to determine the residual cancer burden grade III (RCB-III) after surgery.

The total number of patients to be included in this study is 78 patients.

The duration of the study, from first patient visit to last patient visit will be approximately 90 months (Including follow-ups)

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with histologically confirmed diagnosis of primary unilateral invasive early breast cancer with longest tumor size in breast ≥ 2cm, or < 2 cm with axillary involvement. In case of a multifocal tumor (tumor foci located in the same quadrant) the largest lesion must be ≥ 2cm (unless axillary involvement) and is designated as the "target" lesion for all subsequent tumor evaluations.
2. The breast tumors must be ER positive: more than 1% of stained tumor cells by immuno-histochemistry (IHC), and HER2 negative: 0, or 1+ score by IHC, or 2+ with fluorescence in situ hybridization (FISH)/chromogenic in situ hybridization (CISH) negative for HER2 amplification (defined as a ratio of HER2/neu copies to chromosome 17 centromere (CEP17) signals <1.8), according to the local laboratory).
3. Are clear candidates to receive chemotherapy by the investigator criteria.
4. Are at least 18 years of age.
5. Have at least one unidimensionally measurable lesion by RECIST [65] version 1.1, measured by mammogram.
6. Have adequate performance status: Eastern Cooperative Oncology Group (ECOG) <2
7. Have adequate renal and liver function and bone marrow reserve as follows:

   * Bone marrow: absolute neutrophil count (ANC) > or = 1.500/mm3 (1.5 x 109/L); platelet count > or = 100.000/mm3 (100.0 x 109/L); and hemoglobin > or = 9 g/dL.
   * Hepatic: bilirubin < or = 1.5 times the upper limit of normal (x ULN); alkaline phosphatase (ALP), aspartate transaminase (AST), and alanine transaminase (ALT) < or = 2.5 * ULN and Albumin ≥ 2.5 g/dL.
   * Renal: serum creatinine < 1.5 x ULN.
8. Exhibit patient compliance and geographic proximity that allow for adequate follow-up
9. Entry informed consent form signed by the patient.

Exclusion Criteria:

1. Inflammatory breast cancer (T4d) and supraclavicular lymph nodes (N3)
2. Synchronous contralateral or multicentric breast cancer.
3. Clinical or radiologic evidence of metastatic disease. Chest examination by x-ray or CT-scan, abdominal examination by CT-scan, bone examination by bone scan as well as other radiological methods in case of suspicion must be performed before enrollment in order to rule out metastasis.
4. Second primary malignancy, except adequately treated carcinoma in situ of the cervix, stage I colon cancer, non-invasive melanoma, basal or squamous cell carcinomas of the skin, ipsilateral ductal carcinoma in-situ (DCIS) of the breast and lobular carcinoma in-situ (LCIS) of the breast; unless that prior malignancy was diagnosed and definitively treated more than 5 years ago with no subsequent evidence of recurrence.
5. Prior or concurrent anti-cancer therapy for current disease (hormone therapy, chemotherapy, radiotherapy, immunotherapy, biological therapy other than the trial therapies).
6. Concurrent treatment with any hormonal treatment either for osteoporosis or as replacement therapy.
7. Patients with known hypersensitivity to nab-paclitaxel or any of its components.
8. Previous neuropathy grade >1 according to the NCI-CTCAE vs 4.03 criteria
9. Have received treatment within the last 4 weeks with a drug that has not received regulatory approval for any indication at the time of study entry.
10. Have any serious concomitant systemic disorder incompatible with the study (at the discretion of investigator).
11. Patient is pregnant or breast feeding or planning to become pregnant within the six months after the end of treatment. Women with child-bearing potential must be performed a pregnancy serum or urine testing within 7 days prior to study entry according to institutional standards and should use an adequate non-hormonal contraceptive method (intra-uterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly or surgically sterilized) during treatment with study drugs and within the six months after the end of treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2012-04-17 (Actual); Primary Completion 2014-06-01 (Actual); Study Completion 2018-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hospital General Universitario Gregorio Marañón
Locations (13):
- Spain (13):
  - Corporación Sanitaria Parc Taulí, Sabadell, Barcelona
  - Instituto Oncológico de Guipúzcoa, Donostia / San Sebastian, Guipúzcoa
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Clinic i Provincial, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital La Paz, Madrid
  - Hospital Universitario Morales Meseguer, Murcia
  - Hospital Virgen de la Salud, Toledo
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Miguel Servet, Zaragoza

REFERENCES:
- [Result] Martin M, Chacon JI, Anton A, Plazaola A, Garcia-Martinez E, Segui MA, Sanchez-Rovira P, Palacios J, Calvo L, Esteban C, Espinosa E, Barnadas A, Batista N, Guerrero A, Munoz M, Romio E, Rodriguez-Martin C, Caballero R, Casas MI, Rojo F, Carrasco E, Antolin S. Neoadjuvant Therapy with Weekly Nanoparticle Albumin-Bound Paclitaxel for Luminal Early Breast Cancer Patients: Results from the NABRAX Study (GEICAM/2011-02), a Multicenter, Non-Randomized, Phase II Trial, with a Companion Biomarker Analysis. Oncologist. 2017 Nov;22(11):1301-1308. doi: 10.1634/theoncologist.2017-0052. Epub 2017 Jul 12. PMID 28701571
- See also: Sponsor's web — http://www.geicam.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There are two patients that have not received any cycle and they are excluded of analysis by ITT criterium: One patient did not receive any cycle, ended treatment by investigator´s criterium and the other patient withdrawn informed consent before starting the treatment.
Groups:
- Nab-Paclitaxel: The patients will be included to receive 3 weekly nab-paclitaxel doses of 150 mg/m2 with one week of rest for 4 cycles.
  Nab-paclitaxel
Period: Overall Study
Arm/Group | Nab-Paclitaxel
Started | 83
Completed | 75
Not Completed | 8
Not completed — Physician Decision | 1
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: From the 83 patients registered, there were 2 patients that had not received any cycle and they were excluded of analysis by Intent To Treat (ITT) criterium: One patient did not receive any cycle, ended treatment by investigator´s criterium and the other patient withdrawn informed consent before starting the treatment.
Arm/Group | Nab-Paclitaxel
Number analyzed (Participants) | 81
Age, Continuous [Median (Full Range); unit: years] | 47 [28 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 79
  Hispanic | 2
Menopausal Status [Count of Participants; unit: Participants]
  Premenopausal | 52
  Postmenopausal | 29
Hormonal status [Count of Participants; unit: Participants]
  Estrogen Receptor (ER) (+) and Progesterone R (+) | 62
  ER (+) and Progesterone R (-) | 17
  ER (+) and Progesterone R (Not available) | 2
Eastern Cooperative Oncology Group (ECOG) status [Count of Participants; unit: Participants] — ECOG score runs from 0 to 5, with 0 denoting perfect health and 5 death. ECOG 0: Asymptomatic ECOG 1: Symptomatic but completely ambulatory ECOG 2: Symptomatic, <50% in bed during the day ECOG 3: Symptomatic, >50% in bed, but not bedbound ECOG 4: Bedbound ECOG 5: Death
  Participants
    ECOG 0 | 79
    ECOG 1 | 2
Clinical Tumor size [Count of Participants; unit: Participants] — Tumor (T) size describes the size of the tumour. Larger T is associated with inferior survival.
  TX: can't be assessed. Tis: ductal carcinoma in situ. T1: tumour is 2 centimetres (cm) across or less. T1mi: tumour is 0.1cm across or less T1a: tumour >0.1 cm but <0.5 cm T1b: tumour >0.5 cm but <1 cm T1c: tumour >1 cm but <2 cm T2: tumour >2 cm but <5 cm across T3: tumour >5 cm across T4a: tumour has spread into the chest wall T4b: tumour has spread into the skin and the breast might be swollen T4c: tumour has spread to both the skin and the chest wall T4d: inflammatory carcinoma
  Participants
    T1 | 9
    T1c | 8
    T2 | 42
    T3 | 18
    T4a | 1
    T4b | 3
Clinical Nodal status [Count of Participants; unit: Participants] — Node (N) describes whether the cancer has spread to the Lymph Nodes (LN). Prognosis is better when cancer has not spread to the LN. The more LN that contain cancer, the poorer prognosis tends to be.
  NX: LN can't be assessed N0: no Cancer Cells (CC) N1: CC in the LN in the armpit but the nodes are not stuck to surrounding tissues.
  N2a: CC in the LN in the armpit, which are stuck to each other and to other structures.
  N2b: CC in the LN behind the breast bone. N3a: CC in LN below the collarbone. N3b: CC in LN in the armpit and behind the breastbone.
  Participants
    N0 | 30
    N1 | 43
    N2 | 5
    NX | 3
Clinical Stage [Count of Participants; unit: Participants] — Clinical Stages:
  Stage 0: Abnormal cells are present but have not spread to nearby tissue. Also called carcinoma in situ (CIS). CIS is not cancer, but it may become cancer.
  Stage I, Stage II, and Stage III: Cancer is present. The higher the number, the larger the cancer tumor and the more it has spread into nearby tissues.
  Stage IV: The cancer has spread to distant parts of the body.
  Participants
    Stage I | 4
    Stage II | 56
    Stage III | 18
    Unknown | 3
Histopathologic Grade [Count of Participants; unit: Participants] — Cancer cells are given a Grade (G) when they are removed from the breast and checked under a microscope. The G is based on how much the cancer cells look like normal cells.
  G1 or well differentiated (score 3, 4, or 5): cells are slower-growing, and look more like normal breast tissue.
  G2 or moderately differentiated (score 6, 7): cells are growing at a speed of and look like cells somewhere between G1 and 3.
  G3 or poorly differentiated (score 8, 9): cells look very different from normal and will probably grow and spread faster.
  Participants
    Grade 1 | 9
    Grade 2 | 39
    Grade 3 | 26
    Unknown | 7
Breast Surgery Planned [Count of Participants; unit: Participants]
  Mastectomy | 50
  Quadrantectomy | 17
  Lumpectomy | 10
  Not available | 4

OUTCOME MEASURES:

1. Primary Outcome: The Residual Cancer Burden Grade III (RCB-III).
Description: The RCB-III was reported, including a 95% confidence interval. The estimate of the RCB-III was calculated as follows:
  Overall Response Rate = Number of patients with RCB-III / Intent to treat (ITT) population
Time Frame: After surgery, up to 4 months
Population: From the 83 patients registered, there were 2 patients that had not received any cycle and they were excluded of analysis by Intent To Treat (ITT) criterium: One patient did not receive any cycle, ended treatment by investigator´s criterium and the other patient withdrawn informed consent before starting the treatment.
  Unknown: The RCB evaluation was available for 80 of the 81 treated patients (one patient received three cycles but refused further treatment and withdrew the informed consent).
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-Paclitaxel
Number analyzed (Participants) | 81
Participants
  RCB III: Extensive residual disease (>3.28) | 23
  RCB II: Moderate residual disease (1.36-3.28) | 37
  RCB I: Minimal residual disease (>0-1.36) | 14
  RCB 0: No residual disease (0) | 6
  Unknown | 1

2. Secondary Outcome: Pathologic Complete Response (pCR) Rate
Description: Objective Response was measured following the Response Evaluation Criteria In Solid Tumors (RECIST 1.1) criteria. For the purpose of this study a response is defined as the achievement of a complete or partial response measured by breast MRI.
  Pathological complete response (pCR) was evaluated following the Symmans method at the time of the definitive surgery. For the purpose of this study RCB-0 was considered a pCR.
  The pCR (RCB-0) rate (pCRR) was reported including a 95% confidence interval. The estimate of the pCR rate was calculated as follows by central laboratory:
  pCR Rate = Number of patients with pCR / ITT population.
Time Frame: After surgery, up to 4 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-Paclitaxel
Number analyzed (Participants) | 81
Participants | 6

3. Secondary Outcome: Objective Response Rate (ORR) by Magnetic Resonance Imaging (MRI)
Description: The ORR was reported including a 95% confidence interval. The estimate of the ORR was determined according to RECIST 1.1 and measured by MRI and mammogram in patients treated with this regimen. ORR was calculated as follows:
  Overall Response Rate = Number of Complete Responses (CRs), Partial Responses (PRs) / ITT population
Time Frame: After surgery, up to 4 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-Paclitaxel
Number analyzed (Participants) | 81
Participants | 62

4. Secondary Outcome: Objective Response Rate (ORR) by Mammogram
Description: The ORR was reported including a 95% confidence interval. The estimate of the ORR was determined according to RECIST 1.1 and measured by MRI and mammogram in patients treated with this regimen. ORR was calculated as follows:
  Overall Response Rate = Number of CRs, PRs / ITT population
Time Frame: After surgery, up to 4 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-Paclitaxel
Number analyzed (Participants) | 81
Participants | 49

5. Secondary Outcome: Invasive Disease Free Survival (IDFS)
Description: IDFS was defined as the time (days) from the date of randomization until the date of objective recurrent disease (local, regional or distant), second primary invasive malignancy (breast or non-breast) or death from any cause. For patients not known to have died as of the data cut-off date and who do not have recurrent disease or second primary tumor, invasive disease-free survival will be censored at the last contact date. Ductal carcinoma in-situ (DCIS) will not be considered an event for the purpose of this analysis.
Time Frame: Up to 6 years
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Nab-Paclitaxel
Number analyzed (Participants) | 81
years | 4.89 (1.10)

6. Secondary Outcome: Rate of Conversion to Breast Conserving Surgery (BCS)
Description: The conversion from the initially planned mastectomy to BCS was reported including a 95% confidence interval. The estimate of the rate of conversion to BCS was calculated as follows:
  BCS rate = Number of patients with BCS / Number of patients with initially planned mastectomy.
Time Frame: After surgery, up to 4 months
Population: From the 83 patients registered, there were 2 patients that had not received any cycle and they were excluded of analysis by Intent To Treat (ITT) criterium: One patient did not receive any cycle, ended treatment by investigator´s criterium and the other patient withdrawn informed consent before starting the treatment.
  Mastectomy was de initial planned surgery for 50 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-Paclitaxel
Number analyzed (Participants) | 50
Participants
  Breast-conserving surgery | 20
  No Breast-conserving surgery | 30

7. Secondary Outcome: The Number of Participants Who Experienced Adverse Events (AE)
Description: Incidence of adverse events by maximum CTCAE grade (v4.03; NCI 2010) that occur during the study treatment period or within 30 days of the last dose of study treatment, regardless of causality and according to the relationship to study drug as assessed by the investigator, were collected and evaluated.
Time Frame: During treatment and until 30 days after the last dose of each patient study treatment
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-Paclitaxel
Number analyzed (Participants) | 81
Participants | 81

8. Secondary Outcome: Ki67 in Pre-treatment Tumor Samples as Tumor Predictive Marker of Nab-paclitaxel Response
Description: Ki67 was analysed by immunohistochemistry following the American Society of Clinical Oncology and the College of American Pathologists guidelines. The cut-off considered for Ki67 expression was 20% of positively stained tumor cells.
Time Frame: Baseline visit
Population: Of the 81 patients, 77 had available pretreatment tumors for biomarker central analysis. Of these 77, 5 were excluded (3 due to Triple Negative (TN) phenotype, 1 due to missing pathological response data, and 1 due to incomplete central biomarker data). Ki67 was determined in 72 tumors and correlated to RCB (DOI: 10.1634/theoncologist.2017-0052)
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-Paclitaxel
Number analyzed (Participants) | 72
Participants
  ≥ 20 % | 40
  < 20 % | 32

9. Secondary Outcome: Caveolin-1 in Pre-treatment Tumor Samples as Tumor Predictive Marker of Nab-paclitaxel Response
Description: Caveolin (Cav)-1 was evaluated in the stroma and its expression was categorized in low, moderate, or high (tertile). The high expression of Cav-1 was considered as positive.
Time Frame: Baseline visit
Population: 83 patients registered, but 2 patients that had not received any cycle and they were excluded of analysis by Intent To Treat (ITT) criterium.
  Of the 81 patients, 77 had available pretreatment tumors for biomarker central analysis. Of these 77, 5 were excluded (3 due to Triple Negative (TN) phenotype, 1 due to missing pathological response data, and 1 due to incomplete central biomarker data). Cav-1 was determined in 72 tumors and correlated to RCB (DOI: 10.1634/theoncologist.2017-0052)
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-Paclitaxel
Number analyzed (Participants) | 72
Participants
  Positive | 19
  Negative | 53

10. Secondary Outcome: Secreted Protein, Acidic, Cysteine-rich (SPARC) in Pre-treatment Tumor Samples as Tumor Predictive Marker of Nab-paclitaxel Response
Description: SPARC was evaluated for both tumor and stroma. Its expression was categorized as negative when the intensity was absent-to-weak (1), or moderate (11)-to-strong (111) with a proportion of stained cells <10%. Immunolabeling was positive if the intensity was moderate (11)-to-strong (111) and the extent of staining was 10%.
Time Frame: Baseline visit
Population: 83 patients registered, but 2 patients that had not received any cycle and they were excluded of analysis by Intent To Treat (ITT) criterium.
  Of the 81 patients, 77 had available pretreatment tumors for biomarker central analysis. Of these 77, 5 were excluded (3 due to Triple Negative (TN) phenotype, 1 due to missing pathological response data, and 1 due to incomplete central biomarker data). SPARC was determined in 72 tumors and correlated to RCB (DOI: 10.1634/theoncologist.2017-0052)
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-Paclitaxel
Number analyzed (Participants) | 72
Participants
  SPARC stroma: Positive | 65
  SPARC stroma: Negative | 7
  SPARC tumor: Positive | 7
  SPARC tumor: Negative | 65

11. Secondary Outcome: Molecular Tumor Subtypes According to St. Gallen Criteria 2013 in Pre-treatment Tumor Samples as Predictive Marker of Nab-paclitaxel Response
Description: Molecular subtypes were classified according to St. Gallen criteria 2013 and Prat et al. into Luminal A (ER+, Progesterone Receptor (PgR) >20%, Human Epidermal growth factor Receptor 2 - (HER2), Ki67 <14%), Luminal B1 (ER+, HER2-, PgR >20% and/or Ki67 <14%), Luminal B2 (ER+, HER2+, any PgR, any Ki67), TN (ER-, PgR-, HER2-), and HER2-enriched (ER-, PgR-, HER2+) subtypes.
Time Frame: Baseline
Population: 83 patients registered, but 2 patients that had not received any cycle and they were excluded of analysis by Intent To Treat (ITT) criterium.
  Of the 81 patients, 77 had available pretreatment tumors for biomarker central analysis. Of these 77, 5 were excluded (3 due to TN phenotype, 1 due to missing pathological response data, and 1 due to incomplete central biomarker data). Molecular subtypes was determined in 72 tumors and correlated to RCB (DOI: 10.1634/theoncologist.2017-0052)
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-Paclitaxel
Number analyzed (Participants) | 72
Participants
  Luminal A | 19
  Luminal B1 | 53

ADVERSE EVENTS:
Time Frame: All AEs occurring during the study and until the treatment discontinuation visit 30 days after the last study medication, an average of 4 months per participant
Description: From the 83 patients registered, there were 2 patients that had not received any cycle and they were excluded of analysis by Intent To Treat (ITT) criterium: One patient did not receive any cycle, ended treatment by investigator´s criterium and the other patient withdrawn informed consent before starting the treatment.
Arm/Group | Nab-Paclitaxel
All-Cause Mortality (participants affected / at risk) | 4/81
Serious Adverse Events (participants affected / at risk) | 6/81
Other Adverse Events (participants affected / at risk) | 81/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nab-Paclitaxel (N=81)
Community-acquired pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1 — Grade 2
Multiple Sclerosis Relapse (Nervous system disorders) | 1
Local Infection Reservoir Area (Skin and subcutaneous tissue disorders) | 1
Neurotoxicity (Nervous system disorders) | 2 — Grade 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nab-Paclitaxel (N=81)
Neutrophil Count Decreased (Investigations) | 3 — Grade 4
Neutrophil Count Decreased (Investigations) | 10 — Grade 3
Neutrophil count decreased (Investigations) | 22 — Grade 2
Neutrophil Count Decreased (Investigations) | 21 — Grade 1
Hypertension (Vascular disorders) | 6 — Grade 3
Hypertension (Vascular disorders) | 14 — Grade 2
Hypertension (Vascular disorders) | 6 — Grade 1
Alopecia (Skin and subcutaneous tissue disorders) | 54 — Grade 2
Alopecia (Skin and subcutaneous tissue disorders) | 12 — Grade 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 — Grade 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 — Grade 1
Fatigue (General disorders) | 3 — Grade 3
Fatigue (General disorders) | 19 — Grade 2
Fatigue (General disorders) | 39 — Grade 1
Irregular Menstruation (Reproductive system and breast disorders) | 10 — Grade 2
Irregular Menstruation (Reproductive system and breast disorders) | 4 — Grade 1
Myalgia (Musculoskeletal and connective tissue disorders) | 7 — Grade 2
Myalgia (Musculoskeletal and connective tissue disorders) | 15 — Grade 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 22 — Grade 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 40 — Grade 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 — Grade 3
Upper Respiratory Infection (Infections and infestations) | 1 — Grade 3
Upper Respiratory Infection (Infections and infestations) | 6 — Grade 2
Upper Respiratory Infection (Infections and infestations) | 4 — Grade 1
White Blood Cell Decreased (Investigations) | 3 — Grade 3
White Blood Cell Decreased (Investigations) | 21 — Grade 2
White Blood Cell Decreased (Investigations) | 29 — Grade 1
Alanine Aminotransferase Increased (Investigations) | 30 — Grade 1
Aspartate Aminotransferase Increased (Investigations) | 13 — Grade 1
Anemia (Blood and lymphatic system disorders) | 58 — Grade 1
Diarrhea (Gastrointestinal disorders) | 23 — Grade 1
Hyperglycemia (Metabolism and nutrition disorders) | 17 — Grade 1
Mucositis Oral (Gastrointestinal disorders) | 13 — Grade 1
Nausea (Gastrointestinal disorders) | 23 — Grade 1
Nail Changes (Skin and subcutaneous tissue disorders) | 12 — Grade 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less